

#### RESEARCH SUBJECT CONSENT FORM

TITLE: Comparative effectiveness of two acellular matrices products

(DermaCell vs Integra) for management of deep diabetic foot

ulcers - A randomized clinical trial

**PROTOCOL NO.:** None

WIRB® Protocol #20172895

**SPONSOR:** LifeNet Health

**INVESTIGATOR:** Bijan Najafi, PhD

One Baylor Plaza, MS: BCM390 7200 Cambridge St Rm B01.529

Houston, TX, 77030

**United States** 

STUDY-RELATED

**PHONE NUMBER(S):** Bijan Najafi, Ph

713-798-7536

Ivan Marin

713-798-7538 (24 hours)

SUB-

**INVESTIGATOR(S):** Miguel Montero, MD

Joseph Mills, MD Brian Lepow, DPM Jeffrey Ross, DPM, MD

**STUDY** 

**COORDINATOR(S):** Ivan Marin, BS

Louie Morsy, BS

You are being invited to take part in a research study. A person who takes part in a research study is called a research subject, or research participant.

#### What should I know about this research?

- Someone will explain this research to you.
- This form sums up that explanation.
- Taking part in this research is voluntary. Whether you take part is up to you.
- You can choose not to take part. There will be no penalty or loss of benefits to which you are otherwise entitled.
- You can agree to take part and later change your mind. There will be no penalty or loss of benefits to which you are otherwise entitled.
- If you don't understand, ask questions.
- Ask all the questions you want before you decide.

#### Why is this research being done?

The purpose of this research is to compare two different standard of care treatment for deep wounds in feet or lower limbs. We will be testing two different wound products (dermal matrices to assist with healing in case of major tissue loss), DermACell (LifeNet Health, VA) and Bilayer Matrix Wound Dressing (Integra LifeScience, NJ) by placing it in your wound and observing how it improves for each treatment.

You may qualify to participate in this study because you have a deep wound or significant tissue destruction in your feet or legs and your physician would like to apply a dermal product to help heal your wound. Without applying a dermal product, restoring your tissue loss and thus successful healing your wound would be difficult. Both wound products indicated above are considered as standard of care for your wound condition. However, to date, it is not clear which product is better than the other. The purpose of this research is to compare the treatment benefit of one product compared to the other one.

About 50 subjects will take part in this research.

# How long will I be in this research?

We expect that your taking part in this research will last up to 16 weeks. You may also finish the study early, if your wound closes before the 16 weeks are completed. We may interview you by phone or review your health record up to six months post intervention to find out about outcomes of therapy including success or failure of closing your wound. However, no in person visit is necessary.

| Phone number: |
|----------------|
| _ |
| Email address: |

# What happens to me if I agree to take part in this research?

The research study will be conducted at the following locations: Baylor College of Medicine and Baylor St. Luke's Medical Center (BSLMC).

There are a minimum of 17 study related visits for the completion of this study. Each visit will follow your normal appointments with your doctor and the research team will do some tests and

ask questions regarding your health and your wound. Every visit with their tests are described below. You will be put into a study group by chance (like coin toss) at the beginning of the study. Half the participants will be placed in one group and half in the other group. You cannot choose your study group.

During your treatment day, the clinical staff will consent you for your treatment and include all the benefits and risks information of the matrix that will be applied to your wound (either DermACELL or Bilayer Matrix Wound Dressing).

At each study visit, the research staff will complete the procedures in the following order

- 1) Questionnaires
- 2) Wound Care
- 3) Vascular Assessments
- 4) All other procedures

Please see below all questionnaires that will be asked from you.

**Medical History:** The presence of diabetes will be based on American Diabetes Association criteria. This will include: duration and type of diabetes, type of diabetes medication (insulin, oral, combination therapy, diet), previous history of foot ulcers, amputation (toe, foot), lower extremity bypass, lower extremity angioplasty, Coronary artery bypass surgery, cardiac angioplasty, arthritis, liver disease, osteoporosis (bone density), and bone tumors. We will use the Kaplan co-morbidity index to record these disease severities. We will measure height and weight to determine body mass index (BMI). We will evaluate and/or record some of your blood work (only if it is available per your standard of care). These results will be obtained from your medical record at screening/baseline visit.

**Social and Economic Factors:** We will evaluate the following factors: marital status, years of education, type of work, tobacco history (pack years, current smoker, current use of chewing tobacco, previous smoker, no tobacco history), drug history (current, previous history, no drug history), and alcohol history. These factors will be collected at screening/baseline visit. Also, we will collect cost information for your treatment up to 6 months after you enroll in the study.

**Questionnaires:** Quality of Life, Frailty Status, Sleep Quality, Cognitive Status and Device Acceptability: To evaluate functional status we will use well-accepted questionnaires, SF-12 for Quality of Life, Sleep Quality questionnaire (PSQI), MOCA and TSFI for frailty status. In addition, at each visit, we will interview you about your concern with your wound and product (e.g. wound drainage, smell, pain, lack of comfort, etc.), use of any medications for pain or sleeping, the cost of your transport to the clinic, any adverse events (e.g. infection, need to visit a specialist, etc), etc. To see the timeline for each questionnaire, please refer the table below.

**Pain Intensity Assessment (VAS):** You will be provided with a numerical pain scale where you will report your pain intensity. Research staff will document your pain level. (Measurements will be done at every visit).

**Adverse Event Reporting:** Research Staff will document and report any study/non study related incident as per institution regulations. (Measurement will be done at every visit after baseline.)

**Device Acceptability Questionnaire:** You will be handed a questionnaire to evaluate the study device and provide feedback to the research team. We will be asking about your level of satisfaction with product. These may be questions about the time spent to apply the product, the level of comfort, appearance of the product, the appearance of your healed wound (e.g. presence of scarring), ease of walking or standing with the product and after healing, etc. (Measurement will be done at Visit 8 and Visit 16 or your last visit, whichever comes first.)

After, the research staff and physician will evaluate you blood flow and wound with the following procedures:

**Matrix Application:** During your wound treatment (either in operation room or outpatient clinic), your physician will apply the dermal matrix from the group you were placed. The researchers will write down the duration needed for full application of the product. For accurate estimation of time needed for preparation and application, the whole process may be video-recorded for offline estimate of each time.

Vascular Assessment: We will assess quality of your blood flow to your feet using established methods. (Measurements will be done at screening/baseline and visit 16). For this purpose, blood pressure and pulse at your ankle, and arm will be measured using standard devices named SensiLase system (Väsamed) and Doppler Ultrasound Ankle Brachial Index (ABI). In addition, we may use an imaging technique (SPY or Luna, Novadaq) for an accurate assessment of your skin perfusion. For this purpose a fluorescent agent may be injected into your body to allow us observe the blood circulation to your wound. This assessment is optional. If we decided to use imaging method to assess your skin perfusion, the following steps will be done by the Medical/Research staff:

- 1. Ask you to lie flat and comfortably
- 2. Inject the dye/fluorescent agent into your vessels
- 3. Place the Camera above your wound
- 4. Observe your perfusion and blood flow on the monitor of the imaging system and record any notes made by your physician

Indocyanine Green Fluorescence Imaging (SPY or Luna) may be performed based on the medical judgment of your physician. Highly qualified medical/clinical staff will perform this measurement. If so, measurements will take place only during your baseline and treatment day.

**Ankle-Brachial Index:** This test is to measure blood pressure of your ankle and arm while you are at rest. (Measurements will be done on screening/baseline visit and visits 2 & 4).

#### Research Staff will:

- 1. Attach correct sized cuff on ankle and arm.
- 2. Place Doppler probe on your ankle and arm.

- 3. Inflate cuffs above your blood pressure.
- 4. Deflate the cuffs.
- 5. Document values in your records.
- 6. Remove the cuffs from your ankle and arm.

**Skin Perfusion Pressure:** This test will help your physician and researchers know if your tiny blood vessels in your feet are blocked, damaged or if your wound is getting enough blood to heal properly. (Measurements will be done on screening/baseline visit and visits 2 & 4.)

#### Research Staff will:

- 1. Ask you to lie flat.
- 2. Place correct sized pressure cuffs around your ankles.
- 3. Place an adhesive pad along with a sensor as (sensors will not be touching your skin directly) it will measure your Skin Perfusion.
- 4. Inflate the cuffs above your blood pressure.
- 5. Document values in your records.
- 6. Remove cuffs from your ankle.

**Wound Photo:** At every visit, the Medical/Research staff using a standard digital camera will take a digital photo of your wound.

**Wound Assessment:** Evaluations will be based on data collected from wound assessments and photographs. We use acetate tracings and digital photos. Additionally, we will use thermal imaging to track inflammation. (Measurements will be performed at baseline, visit 8, 10, 12, 14 and 16).

**Wound photo:** A digital photo/video will be taken to record wound size reduction. (Measurement will be performed at every visit.)

**Thermal Image:** A thermal camera will be used to obtain an image of your wound and observe swelling.

**Wifi Wound Classification:** Podiatric (foot) physician or vascular surgeon will evaluate the health and wellness of your feet in compliance of standard of care. (Measurement will be done at baseline, visit 8 and 16).

**Granulation Assessment:** Your physician will be looking at how your wound heals. Specifically, they will look at the reddish tissue developing on your wound. A digital photograph will be taken and comments made by your physician will be recorded. (Measurement will be done at visit 6, 7 & 8).

**Wound Care:** Your physician will schedule regular visits after your surgery to provide care to your wound as according to standard of care.

**Dressing Change:** Medical and/or clinical staff will change your dressing weekly or as needed.

**Neuropathy Assessment:** We will use Vibration Perception Threshold (VPT) testing to assess neuropathy. We will place a vibration knob on different regions of your feet to measure your loss of sensation. (Measurements will be done on screening/baseline visit.)

**Upper Extremity Assessment:** Investigators will measure your arm motion using wearable sensors (LegSys). One sensor will be placed around your wrist and another around your elbow. While being at a comfortable position, you will be asked to flex and extend their arm for 20 seconds at a fast speed. You will also be asked to repeat this task but counting backwards as you flex and extend their arm (dual task). (Measurement will be done at baseline, visit 8 and 16.)

Optional Assessments – These may occur at any visit. However, the do not need to performed. Physical Exam: If you are able to stand and walk, the research staff will place 5 sensors named Legsys and Balanses (one on lower back, two on each upper thigh, and two on each shin) attached with elastic straps to test balance and record your walking patterns. Research staff will ensure that the straps are not too tight to avoid poor circulation.

**Physical activity:** If you are able to stand and walk, the research staff will provide you with a small sensor (Pamsys) that will be measuring your physical activity for 48 hours. It will record your number of steps taken, duration of sitting, standing, walking, and lying. It will also record the number of transitions you made from sitting to standing and vice versa. At the end of the visit, you will be given the sensor, which will be worn, around your neck like a pendant. Researchers will provide you with a pre-paid envelope where you may place the device and send it back to the investigating team after 48 hours.

**Heart Rate Monitoring:** A comfortable chest worn sensor (Zephyr BioHarness, Medtronic or BioStamp RC, MC10) will be used to measure physiological signs such as heart rate, skin temperature, and physical activity. This device will be comfortable placed on your chest attached either with two sticky electrodes or with elastic straps if you have sensitive skin. Researchers will attach this device on you for the duration of the visit or during 24 hours.

Now, please read very carefully the description of every visit. All procedures were described above

#### Screening/Baseline Visit \*duration of visit 90 minutes

This visit will take place at Baylor St. Lukes Medical Center during your surgery day. The research staff will perform as described above: Medical History, Questionnaires (Pain, Social Factors, and Quality of Life, Sleep Quality, Cognitive Assessment, Frailty), Matrix application, Upper Extremity Test, Peripheral Neuropathy, Thermal Image, Vascular Assessment, Wound Assessment, Wifi Wound Classification, and Wound photo.

#### Visit 1, 1<sup>st</sup> Follow Up \*duration 50 minutes

This visit will take place at Baylor Clinic for a regular follow up appointment. The research staff will perform as described above: Pain Questionnaire, Adverse Event Reporting, Dressing Change, Wound Photo, and Wound Care.

#### Visit 2, 2<sup>nd</sup> Follow Up \*duration of visit 70 minutes

This visit will take place at Baylor Clinic for a regular follow up appointment. The research staff will perform as described above: Adverse Event Reporting, Wound Assessment, Thermal Image, Dressing Change, Wound Photo, and Wound Care.

## Visit 3, 3<sup>rd</sup> Follow Up \*duration 50 minutes

This visit will take place at Baylor Clinic for a regular follow up appointment. The research staff will perform as described above: Adverse Event Reporting, Dressing Change, Wound Photo, and Wound Care.

# Visit 4, 4<sup>th</sup> Follow Up \*duration of visit 70 minutes

This visit will take place at Baylor Clinic for a regular follow up appointment. The research staff will perform as described above: Pain Questionnaire, Adverse Event Reporting, Sleep Quality Questionnaire, Wound Assessment, Dressing Change, Wound Photo, Thermal Image, and Wound Care.

# Visit 5, 5<sup>th</sup> Follow Up \*duration 70 minutes

This visit will take place at Baylor Clinic for a regular follow up appointment. The research staff will perform as described above: Adverse Event Reporting, Dressing Change, Wound Photo, Granulation Assessment, and Wound Care.

#### Visit 6, 6<sup>th</sup> Follow Up \*duration 70 minutes

This visit will take place at Baylor Clinic for a regular follow up appointment. The research staff will perform as described above: Adverse Event Reporting, Dressing Change, Thermal Image, Wound Photo, Granulation Assessment, and Wound Care.

#### Visit 7, 7<sup>th</sup> Follow Up \*duration 70 minutes

This visit will take place at Baylor Clinic for a regular follow up appointment. The research staff will perform as described above: Adverse Event Reporting, Dressing Change, Wound Photo, Granulation Assessment, and Wound Care.

#### Visit 8, 8<sup>th</sup> Follow Up \*duration 90 minutes

This visit will take place at Baylor Clinic for a regular follow up appointment. The research staff will perform as described above: Pain Questionnaire, Sleep Quality Questionnaire, Device Acceptability Questionnaire, Adverse Event Reporting, Dressing Change, Wound Photo, Wound Assessment, Granulation Assessment, Wound Care, Wifi Wound Classification, Thermal Image, and Upper Extremity Assessment.

# Visit 9, 9th Follow Up \*duration 40 minutes

This visit will take place at Baylor Clinic for a study-only follow up appointment. The research staff will perform as described above: Adverse Event Reporting, Dressing Change, Wound Photo.

#### Visit 10, 10<sup>th</sup> Follow Up \*duration 70

This visit will take place at Baylor Clinic for a regular follow up appointment. The research staff will perform as described above: Adverse Event Reporting, Dressing Change, Thermal Image, Wound Photo, Wound Care, Wound Assessment.

# Visit 11, 11<sup>th</sup> Follow Up \*duration 40 minutes

This visit will take place at Baylor Clinic for a study-only follow up appointment. The research staff will perform as described above: Adverse Event Reporting, Dressing Change, Wound Photo.

# Visit 12, 12<sup>th</sup> Follow Up \*duration 75 minutes

This visit will take place at Baylor Clinic for a regular follow up appointment. The research staff will perform as described above: Pain Questionnaire, Sleep Quality Questionnaire, Adverse Event Reporting, Dressing Change, Wound Photo, Wound Assessment, Thermal Image, Wound Care.

# Visit 13, 13<sup>th</sup> Follow Up \*duration 40 minutes

This visit will take place at Baylor Clinic for a study-only follow up appointment. The research staff will perform as described above: Adverse Event Reporting, Dressing Change, Wound Photo.

#### Visit 14, 14<sup>th</sup> Follow Up \*duration 70 minutes

This visit will take place at Baylor Clinic for a regular follow up appointment. The research staff will perform as described above: Adverse Event Reporting, Dressing Change, Thermal Image, Wound Photo, Wound Care, Wound Assessment.

#### Visit 15, 15<sup>th</sup> Follow Up \*duration 40 minutes

This visit will take place at Baylor Clinic for a study-only follow up appointment. The research staff will perform as described above: Adverse Event Reporting, Dressing Change, Wound Photo.

#### Visit 16, 16<sup>th</sup> Follow up, OR Last Visit \*duration 90 minutes

This visit will take place at Baylor Clinic for a regular follow up appointment. The research staff will perform as described above. Pain Questionnaire. Sleep Quality Questionnaire. Device

| Acceptability Questionnaire, Adverse Event Reporting, Dressing Change, Wound Photo, Chermal Image, Wound Assessment, Vascular Assessment, Granulation Assessment, Wound Care, Wifi Wound Classification, Upper Extremity Assessment. | l |
|---|---|
| Please provide your Emergency Contact information: | |
| Contact name: | |
| Relationship: | |
| Phone number: | |

| The researchers will take digital photographs and videotape of you during the study. This is done |
|---|
| using a normal camera. The images and videos may be presented in scientific presentations and |
| scientific papers. Your photos and videos will not be used for commercial or marketing purpose. |

| I agree to have my photographs/videotape used and presented in scientific presentation or scientific publication. |
|---|
| I do NOT agree to have my photographs/videotape used and presented in scientific presentation or scientific publication. |
| If you are eligible, the research personnel would like to contact you in the future for participation in other research studies. You are not required to participate in these studies and your medical care or involvement with the current research study will in no way be affected if you choose not to participate. You may ask us to stop contacting you at any time. |
| I agree to be contacted for future research studies. |

The research personnel may call you during your participation in the study with any study-related questions.

I do not agree to be contacted for future research studies.

| Visit | Baseline | Application | | | | | | | | F | ollo | w-up | ) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| # | 0 | 7.66 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |
| Consent | X | | | | | | | | | | | | | | | | | |
| Screening | Х | | | | | | | | | | | | | | | | | |
| Medical<br>History | Х | | | | | | | | | | | | | | | | | |
| Neuropathy<br>Assessment | X | | | | | | | | | | | | | | | | | |
| Dermal matrix application | | X | | | | | | | | | | | | | | | | |
| Dressing changes | | | Х | Х | Х | Х | X | X | Х | Х | Х | Х | X | Х | Х | Х | Х | X |
| Granulation assessment | | | | | | | | X | X | X | | | | | | | | |
| Wound<br>Assessment | Х | | | | | | | | | Х | | X | | X | | X | | Х |
| WiFi wound classification | Х | | | | | | | | | Х | | | | | | | | X |
| Vascular<br>Assessments | Х | | | | | | | | | | | | | | | | | X |
| Wound Photos | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Thermal<br>Images | Х | | | X | | Х | | Х | | Х | | Х | | X | | Х | | Х |
| Wound Care<br>(standard of<br>care) | Х | | Х | Х | X | Х | X | Х | X | Х | | Х | | Х | | Х | | Х |
| Optional assessments | | | X | X | X | X | X | X | X | X | X | X | X | X | Х | X | X | X |

| Adverse<br>Events<br>Reporting | Х | Х | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Pain questionnaires and patient-centered outcomes | Х | X | | | X | | | | X | | | | X | | | | X |
| Sleep quality index | Х | | | | X | | | | X | | | | X | | | | X |
| Device<br>Acceptability<br>Questionnaire | | | | | | | | | X | | | | | | | | Х |

#### What are my responsibilities if I take part in this research?

If you take part in this research, you will be responsible to: Describe the responsibilities of the subject.

- Follow the instructions that your physician gives your regarding your treatment.
- Come to your study visits.
- Avoid walking long distances.
- Contact the research staff if you have any issues with your treatment or have any adverse events (example, hospitalization).

## Could being in this research hurt me?

The study devices and assessment tools that will be used in the study are non-invasive, safe, non-toxic and do not emit any radiation. However, like any battery-powered system, there is also a minimum risk of device malfunctioning and overheating. Please contact the research staff immediately if you experience overheating or device malfunctioning. In addition, the study devices are not waterproof, and although they use a low powered battery (similar to a cell-phone battery), they should not be submerged in water. If you need to take a shower or going swimming, please remove these devices.

When the research staff provide you with either the Physical Activity Monitor or Heart Rate Monitoring device, please make sure to pay extra attention not to damage or lose the device. However, in situations that the device was damaged for any reason, please notify the research staff at your earliest convenience. You will not be charged for any damage or loss of the device. The device may be replaced upon availability.

A vibration perception device will be used to monitor progress and diagnose severity of DPN in lower extremities. The vibration range will be from 0-50 Volts. You may feel slight discomfort from the vibration. This device is compliant with medical electrical device safety.

There is a risk of interference from the device, which may be used to monitor your heart rate (Zephyr Bioharness) in the functionality of pacemaker/ICD devices. Therefore, if you have pacemaker/ICD please inform study staff to avoid using this device on you.

| Do you | have pacemaker or ICD | device? Please ii | nitial below. |
|--------|-----------------------|-------------------|---------------|
| | YES | | |
| | NO | | |

## Will it cost me money to take part in this research?

Taking part in this research may lead to added costs to you, such as:

There are no additional costs to you associated with taking part in this study. Your insurance will be billed for your regular care (such as debridement) and all other study tests will be billed to the sponsor of the study.

#### Will being in this research benefit me?

We cannot promise any benefits to you or others from your taking part in this research. However, possible benefits to you include faster wound healing. Additionally we hope the information learned from this study will help other people with chronic ulcers.

# What other choices do I have besides taking part in this research? Instead of being in this research, your choices may include:

- You may choose not to participate in the study, and still receive DermACell or Bilayer Matrix Wound Dressing outside the study.
  - Treatment with special dressing and bandages.
  - Treatment with other acellular dermal matrices.

# What happens to the information collected for this research?

Your private information and your medical record will be shared with individuals and organizations that conduct or watch over this research, including:

- The research sponsor
- People who work with the research sponsor
- The Principal Investigator
- Research study staff
- Government agencies, such as the Food and Drug Administration
- The Institutional Review Board (IRB) that reviewed this research

We may publish the results of this research. However, we will keep your name and other identifying information confidential.

We protect your information from disclosure to others to the extent required by law. We cannot promise complete secrecy.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### RESEARCH RELATED HEALTH INFORMATION

If you sign this document, you give permission to people who give medical care and ensure quality from Baylor College of Medicine and Baylor St. Luke's Medical Center to use or disclose (release) your health information that identifies you for the research study described in this document. Your information will be given out for regulatory purposes, to conduct the study, and to help ensure the study was done correctly.

The health information that we may use or disclose (release) for this research includes:

- Information from health records such as diagnoses, progress notes, medications, lab or radiology findings, etc.
- Specific information concerning alcohol abuse
- Specific information concerning drug abuse
- Demographic information (name, D.O.B., age, gender, race, etc.)
- Full Social Security #
- Billing or financial records
- Photographs, videotapes, and/or audiotapes of you

The health information listed above may be used by and or disclosed (released) to the following:

- The study sponsor or its representatives, including companies it hires to provide studyrelated services
- Western Institutional Review Board (WIRB) and its representatives
- Other Institutional Review Boards and/or affiliate institutions where approval must be obtained and its representatives
- Regulatory and Government health agencies (such as the Food and Drug Administration, Department of Health and Human Services etc.) in the US or other countries (e.g. European Medicines Agency)
- Office of Human Research Protections (OHRP)
- Member of the research team
- Researchers at other centers taking part in the study
- Data safety monitoring board/committees that are responsible for the safety of research subjects
- Other health care providers involved in your care
- Hospital or other accrediting agencies
- Data collected during the study may be published and made publicly available. Data may also be shared with other research groups. However, data that could in any way identify you will not be made public or shared.

Baylor College of Medicine and Baylor St. Luke's Medical Center are required by law to protect your health information. By signing this document, you authorize Baylor College of Medicine and Baylor St. Luke's Medical Center to use and/or disclose (release) your health information for this research. Those persons who receive your health information may not be required by Federal privacy laws (such as the Privacy rule) to protect it and may share your information with others without your permission, if permitted by laws governing them.

Please note that the research does not involve treatment. Baylor College of Medicine and Baylor St. Luke's Medical Center may not condition (withhold or refuse) treating you on whether you sign this Authorization.

Please note that you may change your mind and revoke (take back) this Authorization at any time. Even if you revoke this Authorization, researchers, their staff and their collaborators on this research project, the Institutional Review Board, LifeNet Health and their representatives, regulatory agencies such as the U.S. Department of Health and Human Services, FDA, Baylor College of Medicine, data coordinating center, Data and Safety Monitoring Board, and Baylor St. Luke's Medical Center may still use or disclose health information they already have obtained about you as necessary to maintain the integrity or reliability of the current research. If you revoke this Authorization, you may no longer be allowed to participate in the research described in this Authorization.

To revoke this Authorization, you must write to: Bijan Najafi, PhD, One Baylor Plaza, MS: BCM390. 7200 Cambridge St Rm B01.529, Houston, TX, 77030

This authorization does not have an expiration date. If all information that does or can identify you is removed from your health information, the remaining information will no longer be subject to this authorization and may be used or disclosed for other purposes.

No publication or public presentation about the research described above will reveal your identity without another authorization from you.

# Who can answer my questions about this research?

The investigator, Bijan Najafi, and/or someone he appoints in his place, will try to answer all of your questions. If you have questions, complaints, or concerns at any time, or if you need to report an injury related to the research, you may speak with a member of the study staff: Ivan Marin at 713-798-7538 during the day and after hours

This research is being overseen by an Institutional Review Board ("IRB"). An IRB is a group of people who perform independent review of research studies. You may talk to them at (800) 562-4789, help@wirb.com if:

- You have questions, concerns, or complaints that are not being answered by the research team.
- You are not getting answers from the research team.
- You cannot reach the research team

- You want to talk to someone else about the research.
- You have questions about your rights as a research subject.

#### What if I am injured because of taking part in this research?

If you are injured or get sick because of being in this research, call the study doctor immediately. The study doctor will provide emergency medical treatment. Your insurance may be billed for this treatment. The sponsor will pay any charges that are not covered by insurance policy or the government, provided the injury was not due to your underlying illness or condition and was not caused by you or some other third party. No other payment is routinely available from the study doctor or sponsor.

## Can I be removed from this research without my approval?

The person in charge of this research can remove you from this research without your approval. Possible reasons for removal include:

- It is in your best interest
- You have a side effect that requires stopping the research
- You need a treatment not allowed in this research
- The research is canceled by the sponsor
- You are unable to keep your scheduled appointments

We will tell you about any new information that may affect your health, welfare, or choice to stay in this research.

# What happens if I agree to be in this research, but I change my mind later?

If you decide to leave this research, contact the research team so that the investigator can:

- Remove you from the study
- Inform your treating physician that you have been removed from the study
- Report the cause that you decide not to be a part of the research study.

If you decide to leave the research early, there may be risks with this decision. These may include: Describe the adverse consequences.

# Will I be paid for taking part in this research?

For taking part in this research, you may be paid up to a total of \$1,275. Your compensation will be broken down as follows:

- You will be paid \$75 for every visit you complete. There is a total of 17 visits.
- You will be given a debit card called "ClinCard" at the first day of your visit. Each time you complete a visit, the coordinator will load \$75 to your card. Please note that it may take up to 72 hours for the amount to be loaded in the card. The research coordinator will

IRB APPROVED AS MODIFIED Mar 15, 2019

provide you with some instructions and useful information about your card. Your SSN will be requested for the research team to issue the payments.

• The research study will also cover your parking or transportation expenses to go to your research visits.

#### **SUBJECTS RIGHTS:**

Your signature on this consent form means that you have received the information about this study and that you agree to volunteer for this research study.

You will be given a copy of this signed form to keep. You are not giving up any of your rights by signing this form. Even after you have signed this form, you may change your mind at any time. Please contact the study staff if you decide to stop taking part in this study.

If you choose not to take part in the research or if you decide to stop taking part later, your benefits and services will stay the same as before this study was discussed with you. You will not lose these benefits, services, or rights.

Signing this consent form indicates that you have read this consent form (or have had it read to you), that your questions have been answered to your satisfaction, and that you voluntarily agree to participate in this research study. You will receive a copy of this signed consent form.

Your signature documents your permission for you or the individual named below to take part in this research.

| Signature of adult subject capable of | f consent | Date |
|----------------------------------------------|------------|------|
| Printed name of subject | | Date |
| (not required if subject personally provided | d consent) | Date |
| Signature of person obtaining co | nsent | Date |
| W. CC P. II. | | |
| Witness (if applicable) | Date | |
| Translator (if applicable) | <br>Date | |



#### FORMULARIO DE CONSENTIMIENTO PARA EL SUJETO DE UNA INVESTIGACIÓN

**TÍTULO:** Eficacia comparativa de dos productos de matrices acelulares

(DermaCell frente a Integra) para el control de úlceras profundas

del pie diabético. - Ensayo clínico aleatorizado.

N.º DE PROTOCOLO: Ninguno

N.° de protocolo del WIRB® 20172895

**PATROCINADOR:** LifeNet Health

**INVESTIGADOR:** Bijan Najafi, PhD

One Baylor Plaza, MS: BCM390 7200 Cambridge St Rm B01.529

Houston, TX 77030 Estados Unidos

NÚMEROS DE TELÉFONO

**DEL ESTUDIO:** Bijan Najafi, PhD

713-798-7536

Ivan Marin

713-798-7538 (las 24 horas)

**INVESTIGADORES** 

**AUXILIARES:** Miguel Montero, MD

Joseph Mills, MD Brian Lepow, DPM Jeffrey Ross, DPM, MD

**COORDINADORES** 

**DEL ESTUDIO:** Ivan Marin, BS

Louie Morsy, BS

Se lo invita a participar en un estudio de investigación. La persona que participa en un estudio de investigación se llama sujeto de la investigación o participante de la investigación.

#### ¿Qué debo saber sobre esta investigación?

- Alguien le explicará esta investigación.
- En este formulario, se resume esa explicación.
- La participación en esta investigación es voluntaria. Depende de usted si va a participar.
- Puede elegir no participar. No sufrirá ningún castigo ni la pérdida de los beneficios que de otra forma le corresponden.
- Puede aceptar participar y cambiar de opinión más adelante. No sufrirá ningún castigo ni la pérdida de los beneficios que de otra forma le corresponden.
- Si no entiende, haga preguntas.
- Haga todas las preguntas que quiera antes de decidirse.

## ¿Por qué se realiza esta investigación?

El objetivo de esta investigación es comparar dos tratamientos diferentes de atención estándar para heridas profundas en los pies o las extremidades inferiores. Evaluaremos dos productos diferentes para heridas (matrices dérmicas para ayudar en la cicatrización en caso de pérdida importante de tejido), DermACell (LifeNet Health, VA) y Bilayer Matrix Wound Dressing (Integra LifeScience, NJ). Para ello, cada uno se le colocará en la herida y se observará la mejoría de la herida con cada tratamiento.

Es posible que usted reúna los requisitos para participar en este estudio porque tiene una herida profunda o una destrucción importante de tejido en los pies o las piernas, y el médico quisiera aplicarle un producto dérmico para ayudar en la cicatrización de la herida. Sin la aplicación de un producto dérmico, la recuperación del tejido perdido y, en consecuencia, la cicatrización exitosa de la herida resultarían difíciles. Los dos productos para heridas indicados más arriba se consideran atención estándar para el estado de su herida. Sin embargo, hasta la fecha no está claro cuál producto es mejor que el otro. El objetivo de esta investigación es comparar el beneficio del tratamiento con un producto frente al otro.

En esta investigación, participarán alrededor de 50 sujetos.

# ¿Cuánto tiempo participaré en esta investigación?

Esperamos que su participación en esta investigación dure un máximo de 16 semanas. También es posible que usted finalice el estudio de manera anticipada si la herida se cierra antes de completarse las 16 semanas. Podremos entrevistarlo por teléfono o revisar su historia clínica hasta seis meses después de la intervención para conocer los resultados de la terapia, que incluyen el éxito o el fracaso del cierre de la herida. Sin embargo, no es necesario realizar ninguna visita en persona.

| Número de teléfono: _ | |
|------------------------|------------|
| Dirección de correo el | ectrónico: |

### ¿Qué me sucede si acepto participar en esta investigación?

El estudio de investigación se realizará en los siguientes lugares: Baylor College of Medicine y Baylor St. Luke's Medical Center (BSLMC).

Para completar este estudio, debe realizarse un mínimo de 17 visitas relacionadas con el estudio. Cada visita seguirá a las citas normales con el médico, y el equipo de la investigación realizará algunas pruebas y le hará preguntas relacionadas con su salud y la herida. Más adelante se describe cada visita junto con sus pruebas. Se lo colocará en un grupo del estudio al azar (como cuando se arroja una moneda al aire) al comienzo del estudio. Se colocará a la mitad de los participantes en un grupo y a la otra mitad en el otro grupo. Usted no puede elegir el grupo del estudio en el que participará.

Durante el día del tratamiento, el personal clínico le pedirá su consentimiento para el tratamiento, que incluirá toda la información sobre los riesgos y los beneficios de la matriz que se le aplicará en la herida (DermACELL o Bilayer Matrix Wound Dressing).

En cada visita del estudio, el personal de la investigación realizará los procedimientos en el siguiente orden:

- 1) Cuestionarios.
- 2) Cuidado de la herida.
- 3) Evaluaciones vasculares.
- 4) Todos los demás procedimientos.

Consulte más adelante todos los cuestionarios que se le pedirá que responda.

Antecedentes médicos: La presencia de diabetes se basará en los criterios de American Diabetes Association. Estos incluirán: tipo de diabetes y duración, tipo de medicamentos para la diabetes (insulina, orales, terapia combinada, dieta), antecedentes de úlceras del pie, amputación (dedo del pie, pie), *bypass* en las extremidades inferiores, angioplastia en las extremidades inferiores, cirugía de *bypass* en las arterias coronarias, angioplastia cardíaca, artritis, enfermedad hepática, osteoporosis (densidad ósea) y tumores en los huesos. Usaremos el índice de comorbilidad de Kaplan para registrar la gravedad de estas enfermedades. Mediremos la estatura y el peso para determinar el índice de masa corporal (*body mass index*, BMI). Evaluaremos y/o registraremos los resultados de algunos de los análisis de sangre (solo si se encuentran disponibles como parte de su atención estándar). Estos resultados se obtendrán de su historia clínica en la visita de selección/inicial.

**Factores socioeconómicos:** Evaluaremos los siguientes factores: estado civil, años de escolarización, tipo de trabajo, antecedentes de consumo de tabaco (paquetes por año, fumador en la actualidad, uso actual de tabaco para mascar, fumador en el pasado, sin antecedentes de consumo de tabaco), antecedentes de consumo de drogas (en la actualidad, antecedentes, sin antecedentes de consumo de drogas) y antecedentes de consumo de alcohol. Estos factores se obtendrán en la visita de selección/inicial. Además, obtendremos información sobre los costos del tratamiento hasta 6 meses después de su inscripción en el estudio.

Cuestionarios: Calidad de vida, estado de fragilidad, calidad del sueño, estado cognitivo y aceptabilidad del dispositivo: Para evaluar el estado funcional, usaremos cuestionarios convencionales, SF-12 para la calidad de vida, el cuestionario sobre la calidad del sueño (PSQI), MOCA y TSFI para la determinación del estado de fragilidad. Además, en cada visita le haremos una entrevista sobre su preocupación en cuanto a la herida y el producto (por ejemplo, supuración de la herida, olor, dolor, incomodidad, etc.), el uso de medicamentos para el dolor o para dormir, el costo del traslado a la clínica, los eventos adversos (por ejemplo, infección, necesidad de visitar a un especialista, etc.), etc. Consulte la tabla más adelante para ver el cronograma correspondiente a cada cuestionario.

**Evaluación de la intensidad del dolor (VAS):** Se le entregará una escala numérica de dolor en la que deberá comunicar la intensidad del dolor que tiene. El personal de la investigación documentará su nivel de dolor. (Las mediciones se harán en todas las visitas).

Comunicación de eventos adversos: El personal de la investigación documentará y comunicará cualquier incidente relacionado o no con el estudio, según las normativas de la institución. (La medición se hará en todas las visitas después del inicio).

Cuestionario sobre la aceptabilidad del dispositivo: Se le entregará un cuestionario para evaluar el dispositivo del estudio y aportar su opinión al equipo de la investigación. Le preguntaremos sobre su nivel de satisfacción con el producto. Estas pueden ser preguntas sobre el tiempo dedicado a la aplicación del producto, el nivel de comodidad, el aspecto del producto, el aspecto de la herida cicatrizada (por ejemplo, la presencia de cicatrices), la facilidad para caminar o ponerse de pie con el producto y después de la cicatrización, etc. (La medición se hará en la visita 8 y la visita 16 o en la última visita, lo que ocurra primero).

Posteriormente, el médico y el personal de la investigación le evaluarán el flujo de sangre y la herida con los siguientes procedimientos:

**Aplicación de la matriz:** Durante el tratamiento de la herida (en el quirófano o en la clínica ambulatoria), el médico le aplicará la matriz dérmica del grupo en el que se lo colocó. Los investigadores anotarán la duración necesaria de la aplicación del producto en total. Para un cálculo preciso del tiempo necesario para la preparación y la aplicación, es posible que todo el proceso se grabe en video para un cálculo fuera de línea de cada ocasión.

Evaluación vascular: Evaluaremos la calidad del flujo de sangre hacia los pies mediante el uso de métodos establecidos. (Las mediciones se harán en la selección/el inicio y la visita 16). Para ello, se le medirán la presión arterial y el pulso en el tobillo y el brazo con dispositivos estándar llamados sistema SensiLase (Väsamed), y el índice tobillo-braquial (*ankle brachial index*, ABI) mediante ecografía Doppler. Además, es posible que usemos una técnica de obtención de imágenes (SPY o Luna, Novadaq) para una evaluación precisa de la perfusión cutánea. Para ello, es posible que se le inyecte en el cuerpo un agente fluorescente para permitirnos observar la circulación de la sangre hacia la herida. Esta evaluación es opcional. Si decidimos usar un método de obtención de imágenes para evaluar la perfusión cutánea, el personal médico/de la investigación llevará a cabo los siguientes pasos:

- 1. Le pedirá que se acueste de manera cómoda.
- 2. Le inyectará el colorante/agente fluorescente en los vasos.
- 3. Colocará la cámara sobre la herida.
- 4. Observará la perfusión y el flujo de sangre en el monitor del sistema de obtención de imágenes, y registrará las observaciones que realice el médico.

Es posible que se obtengan imágenes por fluorescencia con verde de indocianina (SPY o Luna), según el criterio médico del médico. A esta medición la realizará personal médico/clínico altamente calificado. En ese caso, las mediciones se harán solo durante el inicio y el día del tratamiento.

**Índice tobillo-braquial:** Esta prueba se usa para medir la presión arterial del tobillo y el brazo mientras usted está en reposo. (Las mediciones se harán en la visita de selección/inicial, y las visitas 2 y 4).

El personal de la investigación hará lo siguiente:

- 1. Le colocará el brazalete de tamaño correcto en el tobillo y el brazo.
- 2. Le colocará la sonda Doppler en el tobillo y el brazo.
- 3. Inflará los brazaletes por encima del valor de su presión arterial.
- 4. Desinflará los brazaletes.
- 5. Documentará los valores en sus registros.
- 6. Le retirará los brazaletes del tobillo y el brazo.

**Presión de perfusión cutánea:** Esta prueba ayudará al médico y a los investigadores a saber si los diminutos vasos sanguíneos de los pies están bloqueados o dañados, o si la herida recibe suficiente sangre para cicatrizar de manera adecuada. (Las mediciones se harán en la visita de selección/inicial, y las visitas 2 y 4).

El personal de la investigación hará lo siguiente:

- 1. Le pedirá que se acueste.
- 2. Le colocará los brazaletes para la presión arterial de tamaño correcto alrededor de los tobillos.
- 3. Le colocará una almohadilla adhesiva junto con un sensor (los sensores no estarán en contacto directo con la piel), ya que este le medirá la perfusión cutánea.
- 4. Inflará los brazaletes por encima del valor de su presión arterial.
- 5. Documentará los valores en sus registros.
- 6. Le retirará los brazaletes de los tobillos.

**Fotografía de la herida:** En cada visita, el personal médico/de la investigación tomará una fotografía digital de la herida con una cámara digital estándar.

**Evaluación de la herida:** Las evaluaciones se basarán en los datos obtenidos de las fotografías y las evaluaciones de la herida. Usaremos trazados en películas de acetato y fotografías digitales. Además, usaremos imágenes térmicas para llevar un registro de la inflamación. (Las mediciones se harán en el inicio, y las visitas 8, 10, 12, 14 y 16).

**Fotografía de la herida:** Se obtendrá un video/una fotografía digital para registrar la disminución del tamaño de la herida. (La medición se hará en todas las visitas).

**Imagen térmica:** Se usará una cámara térmica para obtener una imagen de la herida y observar la hinchazón.

Clasificación WIfI (*Wound*, *Ischemia and foot Infection* [herida, isquemia e infección del pie]) de la herida: El médico podólogo (de los pies) o el cirujano vascular evaluarán la salud y el bienestar de los pies, en cumplimiento con la atención estándar. (La medición se hará al inicio, y en las visitas 8 y 16).

**Evaluación del tejido de granulación:** El médico observará cómo cicatriza la herida. Específicamente, observará el tejido rojizo que se desarrolla alrededor de la herida. Se tomará una fotografía digital y se registrarán los comentarios que realice el médico. (La medición se hará en las visitas 6, 7 y 8).

**Cuidado de la herida:** El médico programará visitas periódicas después de la cirugía para proporcionarle el cuidado de la herida, según la atención estándar.

**Cambio del vendaje:** El personal médico y/o clínico le cambiará el vendaje una vez por semana o según sea necesario.

**Evaluación de neuropatía:** Usaremos las pruebas del umbral de percepción vibratoria (*vibration perception threshold*, VPT) para evaluar la neuropatía. Colocaremos una perilla vibratoria en diferentes regiones de los pies para medir la pérdida de sensibilidad. (Las mediciones se harán en la visita de selección/inicial).

Evaluación de las extremidades superiores: Los investigadores medirán la movilidad de los brazos mediante sensores portátiles (LegSys). Un sensor se le colocará alrededor de la muñeca y otro alrededor del codo. Mientras se encuentre en una posición cómoda, se le pedirá que flexione y extienda el brazo rápidamente durante 20 segundos. También se le pedirá que repita esta tarea, pero contando hacia atrás mientras flexiona y extiende el brazo (tarea doble). (La medición se hará al inicio, y en las visitas 8 y 16).

**Evaluaciones opcionales:** Pueden realizarse en cualquier visita. Sin embargo, no es obligatorio realizarlas.

**Exploración física:** Si puede ponerse de pie y caminar, el personal de la investigación le colocará 5 sensores, llamados Legsys y Balanses (uno en la zona lumbar, dos en la parte superior de cada muslo y dos en cada tibia), sujetos con tiras elásticas para evaluar el equilibrio y registrar los patrones de caminata. El personal de la investigación se asegurará de que las tiras no estén muy ajustadas para evitar una mala circulación.

Actividad física: Si puede ponerse de pie y caminar, el personal de la investigación le proporcionará un pequeño sensor (Pamsys) con el que se medirá su actividad física durante 48 horas. Registrará la cantidad de pasos que dé, y el tiempo que esté sentado, de pie, caminando y acostado. También registrará la cantidad de veces que pasa de estar sentado a ponerse de pie y viceversa. Al final de la visita, se le entregará el sensor, que deberá usarse alrededor del cuello como un colgante. Los investigadores le entregarán un sobre con franqueo postal pago, en el que podrá colocar el dispositivo y devolverlo al equipo de la investigación después de las 48 horas.

Control de la frecuencia cardíaca: Se usará un sensor en el pecho que no causa molestias (Zephyr BioHarness, Medtronic o BioStamp RC, MC10) para medir los signos fisiológicos, como la frecuencia cardíaca, la temperatura de la piel y la actividad física. Este dispositivo se le colocará cómodamente en el pecho y se sujetará con dos electrodos adhesivos o con tiras elásticas si tiene la piel sensible. Los investigadores le colocarán este dispositivo todo el tiempo que dure la visita o durante 24 horas.

Ahora, lea con mucha atención la descripción de cada visita. Todos los procedimientos se describieron más arriba.

#### Visita de selección/inicial - \*Duración de la visita: 90 minutos

Esta visita se realizará en Baylor St. Luke's Medical Center durante el día de la cirugía. El personal de la investigación realizará lo siguiente según se describió más arriba: antecedentes médicos, cuestionarios (dolor, factores sociales y calidad de vida, calidad del sueño, evaluación cognitiva, fragilidad), aplicación de la matriz, prueba de las extremidades superiores, neuropatía periférica, imagen térmica, evaluación vascular, evaluación de la herida, clasificación WIfI de la herida y fotografía de la herida.

#### Visita 1, 1.er seguimiento - \*Duración: 50 minutos

Esta visita se realizará en Baylor Clinic durante una cita de seguimiento normal. El personal de la investigación realizará lo siguiente según se describió más arriba: cuestionario sobre el dolor, comunicación de eventos adversos, cambio del vendaje, fotografía de la herida y cuidado de la herida

# Visita 2, 2. do seguimiento - \*Duración de la visita: 70 minutos

Esta visita se realizará en Baylor Clinic durante una cita de seguimiento normal. El personal de la investigación realizará lo siguiente según se describió más arriba: comunicación de eventos adversos, evaluación de la herida, imagen térmica, cambio del vendaje, fotografía de la herida y cuidado de la herida.

<u>Visita 3, 3. er seguimiento - \*Duración: 50 minutos</u> Esta visita se realizará en Baylor Clinic durante una cita de seguimiento normal. El personal de la investigación realizará lo siguiente según se describió más arriba: comunicación de eventos adversos, cambio del vendaje, fotografía de la herida y cuidado de la herida.

#### Visita 4, 4.º seguimiento - \*Duración de la visita: 70 minutos

Esta visita se realizará en Baylor Clinic durante una cita de seguimiento normal. El personal de la investigación realizará lo siguiente según se describió más arriba: cuestionario sobre el dolor, comunicación de eventos adversos, cuestionario sobre la calidad del sueño, evaluación de la herida, cambio del vendaje, fotografía de la herida, imagen térmica y cuidado de la herida.

#### Visita 5, 5.º seguimiento - \*Duración: 70 minutos

Esta visita se realizará en Baylor Clinic durante una cita de seguimiento normal. El personal de la investigación realizará lo siguiente según se describió más arriba: comunicación de eventos adversos, cambio del vendaje, fotografía de la herida, evaluación del tejido de granulación y cuidado de la herida.

#### Visita 6, 6.º seguimiento - \*Duración: 70 minutos

Esta visita se realizará en Baylor Clinic durante una cita de seguimiento normal. El personal de la investigación realizará lo siguiente según se describió más arriba: comunicación de eventos adversos, cambio del vendaje, imagen térmica, fotografía de la herida, evaluación del tejido de granulación y cuidado de la herida.

#### Visita 7, 7.º seguimiento - \*Duración: 70 minutos

Esta visita se realizará en Baylor Clinic durante una cita de seguimiento normal. El personal de la investigación realizará lo siguiente según se describió más arriba: comunicación de eventos adversos, cambio del vendaje, fotografía de la herida, evaluación del tejido de granulación y cuidado de la herida.

#### Visita 8, 8.º seguimiento - \*Duración: 90 minutos

Esta visita se realizará en Baylor Clinic durante una cita de seguimiento normal. El personal de la investigación realizará lo siguiente según se describió más arriba: cuestionario sobre el dolor, cuestionario sobre la calidad del sueño, cuestionario sobre la aceptabilidad del dispositivo, comunicación de eventos adversos, cambio del vendaje, fotografía de la herida, evaluación de la herida, evaluación del tejido de granulación, cuidado de la herida, clasificación WIfI de la herida, imagen térmica y evaluación de las extremidades superiores.

# Visita 9, 9.º seguimiento - \*Duración: 40 minutos

Esta visita se realizará en Baylor Clinic durante una cita de seguimiento exclusiva del estudio. El personal de la investigación realizará lo siguiente según se describió más arriba: comunicación de eventos adversos, cambio del vendaje y fotografía de la herida.

#### Visita 10, 10.º seguimiento - \*Duración: 70 minutos

Esta visita se realizará en Baylor Clinic durante una cita de seguimiento normal. El personal de la investigación realizará lo siguiente según se describió más arriba: comunicación de eventos adversos, cambio del vendaje, imagen térmica, fotografía de la herida, cuidado de la herida y evaluación de la herida.

#### Visita 11, 11. er seguimiento - \*Duración: 40 minutos

Esta visita se realizará en Baylor Clinic durante una cita de seguimiento exclusiva del estudio. El personal de la investigación realizará lo siguiente según se describió más arriba: comunicación de eventos adversos, cambio del vendaje y fotografía de la herida.

# Visita 12, 12. do seguimiento - \*Duración: 75 minutos

Esta visita se realizará en Baylor Clinic durante una cita de seguimiento normal. El personal de la investigación realizará lo siguiente según se describió más arriba: cuestionario sobre el dolor, cuestionario sobre la calidad del sueño, comunicación de eventos adversos, cambio del vendaje, fotografía de la herida, evaluación de la herida, imagen térmica y cuidado de la herida.

#### Visita 13, 13. er seguimiento - \*Duración: 40 minutos

Esta visita se realizará en Baylor Clinic durante una cita de seguimiento exclusiva del estudio. El personal de la investigación realizará lo siguiente según se describió más arriba: comunicación de eventos adversos, cambio del vendaje y fotografía de la herida.

#### Visita 14, 14.º seguimiento - \*Duración: 70 minutos

Esta visita se realizará en Baylor Clinic durante una cita de seguimiento normal. El personal de la investigación realizará lo siguiente según se describió más arriba: comunicación de eventos adversos, cambio del vendaje, imagen térmica, fotografía de la herida, cuidado de la herida y evaluación de la herida.

#### Visita 15, 15.º seguimiento - \*Duración: 40 minutos

Esta visita se realizará en Baylor Clinic durante una cita de seguimiento exclusiva del estudio. El personal de la investigación realizará lo siguiente según se describió más arriba: comunicación de eventos adversos, cambio del vendaje y fotografía de la herida.

#### Visita 16, 16.º seguimiento O visita final - \*Duración: 90 minutos

Esta visita se realizará en Baylor Clinic durante una cita de seguimiento normal. El personal de la investigación realizará lo siguiente según se describió más arriba: cuestionario sobre el dolor, cuestionario sobre la calidad del sueño, cuestionario sobre la aceptabilidad del dispositivo, comunicación de eventos adversos, cambio del vendaje, fotografía de la herida, imagen térmica, evaluación de la herida, evaluación vascular, evaluación del tejido de granulación, cuidado de la herida, clasificación WIfI de la herida y evaluación de las extremidades superiores.

| Nombre del contacto: |
|----------------------|
| Relación: |
| Número de teléfono: |

Proporcione la información de su contacto para emergencias:

| una cáma | as y artículos científicos. Sus fotografías y videos no se usarán con fines comerciales |
|---|---|
| | cámara normal. Es posible que las imágenes y los videos se incluyan en presentaciones ificas y artículos científicos. Sus fotografías y videos no se usarán con fines comerciales promoción comercial. Acepto que mis fotografías/cintas de video se usen y se incluyan en presentaciones científicas o en publicaciones científicas. NO acepto que mis fotografías/cintas de video se usen ni se incluyan en presentaciones científicas ni en publicaciones científicas. apto, el personal de la investigación quisiera comunicarse con usted en el futuro en relación a participación en otros estudios de investigación. No se le exige que participe en estos lios y su atención médica o su participación en el estudio de investigación actual no se verán adas de ninguna manera si elige no participar. Puede pedirnos que dejemos de comunicarnos usted en cualquier momento. Acepto que se comuniquen conmigo en relación con futuros estudios de investigación. No acepto que se comuniquen conmigo en relación con futuros estudios |
| con la pa<br>estudios<br>afectadas | articipación en otros estudios de investigación. No se le exige que participe en estos y su atención médica o su participación en el estudio de investigación actual no se verán se de ninguna manera si elige no participar. Puede pedirnos que dejemos de comunicarnos |
| | Acepto que se comuniquen conmigo en relación con futuros estudios de investigación. |
| | No acepto que se comuniquen conmigo en relación con futuros estudios de investigación. |

El personal de la investigación puede llamarlo durante su participación en el estudio para hacer preguntas relacionadas con el estudio.

| Visita | Inicio | Aplicación | | | | | | | | Seg | juin | nient | to | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N.º | 0 | | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |
| Consentimiento. | Х | | | | | | | | | | | | | | | | | |
| Selección. | X | | | | | | | | | | | | | | | | | |
| Antecedentes médicos. | X | | | | | | | | | | | | | | | | | |
| Evaluación de neuropatía. | X | | | | | | | | | | | | | | | | | |
| Aplicación de la matriz dérmica. | | X | | | | | | | | | | | | | | | | |
| Cambios del vendaje. | | | Х | Х | Х | Х | X | X | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Evaluación del tejido de granulación. | | | | | | | | X | X | X | | | | | | | | |
| Evaluación de la herida. | Х | | | | | | | | | Х | | X | | X | | X | | X |
| Clasificación Wlfl<br>de la herida. | Х | | | | | | | | | Х | | | | | | | | X |
| Evaluaciones vasculares. | Х | | | | | | | | | | | | | | | | | Х |
| Fotografías de la herida. | Х | Х | Х | X | X | X | X | X | X | Х | X | X | Х | X | Х | X | X | Х |
| lmágenes<br>térmicas. | Х | | | X | | Х | | X | | Х | | X | | X | | X | | Х |

| Visita | Inicio | Aplicación | | | | | | | | Seg | juin | nien | to | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Cuidado de la herida (atención estándar). | Х | | X | Х | Х | Х | Х | Х | Х | Х | | X | | Х | | X | | Х |
| Evaluaciones opcionales. | | | X | X | X | | X | X | X | X | X | Х | Х | Х | Х | X | X | X |
| Comunicación de eventos adversos. | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Cuestionarios<br>sobre el dolor y<br>resultados<br>centrados en el<br>paciente. | X | | X | | | X | | | | X | | | | X | | | | X |
| Índice de calidad del sueño. | Х | | | | | X | | | | X | | | | X | | | | X |
| Cuestionario<br>sobre la<br>aceptabilidad del<br>dispositivo. | | | | | | | | | | Х | | | | | | | | X |

# ¿Cuáles son mis responsabilidades si participo en esta investigación?

Si participa en esta investigación, será responsable de: Describir las responsabilidades del sujeto.

- Seguir las instrucciones que le dé el médico respecto del tratamiento.
- Ir a las visitas del estudio.
- Evitar caminar grandes distancias.
- Comunicarse con el personal de la investigación si tiene problemas con el tratamiento o cualquier evento adverso (por ejemplo, hospitalización).

# ¿Podría causarme daño participar en esta investigación?

Los dispositivos del estudio y las herramientas de evaluación que se usarán en el estudio son seguros, no son invasivos ni tóxicos, ni emiten radiación. Sin embargo, como cualquier sistema alimentado por batería, también hay un riesgo mínimo de desperfecto del dispositivo y sobrecalentamiento. Comuníquese de inmediato con el personal de la investigación si se produce sobrecalentamiento o un desperfecto del dispositivo. Además, los dispositivos del estudio no son resistentes al agua, y si bien usan una batería de baja potencia (similar a la batería de un teléfono celular), no deben sumergirse en agua. Si tiene que ducharse o va a nadar, retire estos dispositivos.

Cuando el personal de la investigación le entregue el dispositivo de control de la actividad física o de control de la frecuencia cardíaca, asegúrese de prestar especial atención en no dañarlo ni perderlo. Sin embargo, en situaciones en las que por cualquier motivo el dispositivo se haya dañado, comuníqueselo al personal de la investigación tan pronto como pueda. No tendrá que pagar en caso de daño o pérdida del dispositivo. El dispositivo podrá reemplazarse según su disponibilidad.

Se usará un dispositivo de percepción vibratoria para controlar la evolución y diagnosticar la gravedad de la neuropatía periférica diabética (*diabetic peripheral neuropathy*, DPN) en las extremidades inferiores. La vibración variará de 0 a 50 voltios. Puede sentir molestias leves a causa de la vibración. Este dispositivo cumple con las normas de seguridad de dispositivos médicos eléctricos.

Hay un riesgo de interferencia del dispositivo que puede usarse para controlarle la frecuencia cardíaca (Zephyr Bioharness) en la funcionalidad de marcapasos/dispositivos desfibriladores cardioversores implantables (*implantable cardioverter defibrillators*, ICD). Por lo tanto, si tiene un marcapasos/ICD, comuníqueselo al personal del estudio para evitar el uso de este dispositivo en su caso.

| ¿Tiene un marca | apasos o un dispositiv | vo ICD? Escriba sus | iniciales a continuación | 1. |
|---|---|---|---|---|
| SÍ. | | | | |
| NO. | | | | |

# ¿Me costará dinero participar en esta investigación?

La participación en esta investigación puede generarle costos adicionales a usted, por ejemplo:

No hay ningún costo adicional para usted asociado con la participación en este estudio. Su seguro deberá pagar su atención habitual (como el desbridamiento) y el patrocinador del estudio pagará todas las demás pruebas del estudio.

# ¿Me beneficiará la participación en esta investigación?

No podemos prometer ningún beneficio para usted u otras personas por su participación en esta investigación. Sin embargo, los posibles beneficios para usted incluyen una cicatrización más rápida de la herida. Además, esperamos que la información que se obtenga de este estudio ayude a otras personas con úlceras crónicas.

# ¿Qué otras opciones tengo además de la participación en esta investigación?

En lugar de participar en esta investigación, sus opciones pueden incluir lo siguiente:

- Puede elegir no participar en el estudio e igualmente recibir DermACell o Bilayer Matrix Wound Dressing fuera del estudio.
- Recibir tratamiento con apósitos y vendajes especiales.
- Recibir tratamiento con otras matrices dérmicas acelulares.

# ¿Qué sucede con la información que se reúne para esta investigación?

La información privada sobre usted y su historia clínica se compartirán con personas y organizaciones que realizan o supervisan esta investigación, que incluyen:

- El patrocinador de la investigación.
- Las personas que trabajan con el patrocinador de la investigación.
- El investigador principal.
- El personal del estudio de investigación.
- Las agencias gubernamentales, como la Administración de Alimentos y Medicamentos (*Food and Drug Administration*, FDA).
- El Comité de Revisión Institucional (*Institutional Review Board*, IRB) que revisó esta investigación.

Podemos publicar los resultados de esta investigación. Sin embargo, mantendremos la confidencialidad de su nombre y otra información que lo identifique.

Protegemos la información sobre usted de la entrega a otras personas o entidades en la medida que lo exija la ley. No podemos prometer que se mantenga completamente en secreto.

Según lo exigen las leyes de los EE. UU., se dispondrá de una descripción de este ensayo clínico en http://www.ClinicalTrials.gov. Este sitio web no incluirá información que permita su identificación. A lo sumo, incluirá un resumen de los resultados. Puede consultar este sitio web en cualquier momento.

#### INFORMACIÓN SOBRE LA SALUD RELACIONADA CON LA INVESTIGACIÓN

Si firma este documento, da su permiso para que las personas que brindan atención médica y garantizan la calidad de Baylor College of Medicine y Baylor St. Luke's Medical Center usen o entreguen (revelen) la información sobre su salud que lo identifica para el estudio de investigación que se describe en este documento. La información sobre usted se entregará con objetivos de regulación, para realizar el estudio y para ayudar a garantizar que el estudio se haya realizado correctamente.

La información sobre la salud que podemos usar o entregar (revelar) para esta investigación incluye:

- Información de la historia clínica, como diagnósticos, notas de evolución, medicamentos, datos radiológicos o de laboratorio, etc.
- Información específica sobre alcoholismo.
- Información específica sobre drogadicción.
- Información demográfica (nombre, fecha de nacimiento, edad, sexo, raza, etc.).
- N.º de seguro social completo.
- Registros financieros o de facturación.
- Fotografías, cintas de video y/o cintas de audio de usted.

La información sobre la salud detallada más arriba puede ser usada por las siguientes personas o entidades y/o entregada (revelada) a ellas:

- El patrocinador del estudio o sus representantes, incluidas las compañías contratadas para prestar servicios relacionados con el estudio.
- Western Institutional Review Board (WIRB) y sus representantes.
- Otros Comités de Revisión Institucional y/o instituciones afiliadas cuya aprobación se debe obtener, y sus representantes.
- Las agencias de salud gubernamentales y reguladoras (como la Administración de Alimentos y Medicamentos, el Departamento de Salud y Servicios Sociales [*Department of Health and Human Services*, DHHS], etc.) de los Estados Unidos o de otros países (por ejemplo, la Agencia Europea de Medicamentos [*European Medicines Agency*, EMA]).
- La Oficina de Protección de Seres Humanos que Participan en Investigaciones (*Office of Human Research Protections*, OHRP).
- Un integrante del equipo de la investigación.
- Los investigadores de otros centros que participan en el estudio.
- Los comités de supervisión de seguridad de datos que son responsables de la seguridad de los sujetos de una investigación.
- Otros prestadores de atención médica involucrados en su atención.
- El hospital u otras agencias de acreditación.
- Los datos que se obtengan durante el estudio pueden publicarse y ponerse a disposición del público. Además, es posible que se compartan con otros grupos de investigación. Sin embargo, los datos que pudiesen identificarlo de alguna manera no se pondrán a disposición del público ni se compartirán.

Baylor College of Medicine y Baylor St. Luke's Medical Center están obligados por ley a proteger la información sobre su salud. Al firmar este documento, usted autoriza a Baylor College of Medicine y a Baylor St. Luke's Medical Center a usar y/o entregar (revelar) la información sobre su salud para esta investigación. Es posible que las leyes federales de privacidad (como la norma de privacidad) no exijan a las personas que reciban la información sobre su salud que la protejan y tal vez la compartan con otras personas o entidades sin su permiso, si así se los permiten las leyes por las que se rigen.

Tenga en cuenta que la investigación no incluye tratamiento. Baylor College of Medicine y Baylor St. Luke's Medical Center no pueden condicionar (suspender o negar) el tratamiento que le brinden al hecho de que usted firme esta autorización.

Tenga en cuenta que puede cambiar de opinión y revocar (retirar) esta autorización en cualquier momento. Aunque revoque esta autorización, los investigadores, el personal que trabaja con ellos y sus colaboradores en este proyecto de investigación; el Comité de Revisión Institucional; LifeNet Health y sus representantes; las agencias reguladoras, como el Departamento de Salud y Servicios Sociales de los EE. UU.; la FDA; Baylor College of Medicine; el centro de coordinación de datos; el Comité de Control de la Seguridad y los Datos (*Data and Safety Monitoring Board*, DSMB); y Baylor St. Luke's Medical Center podrán seguir usando o entregando la información sobre su salud que ya hayan obtenido, según sea necesario, para mantener la integridad o la confiabilidad de la investigación actual. Si revoca esta autorización, tal vez ya no se le permita participar en la investigación descrita en ella.

Para revocar esta autorización, debe escribir a: Bijan Najafi, PhD, One Baylor Plaza, MS: BCM390, 7200 Cambridge St Rm B01.529, Houston, TX 77030.

Esta autorización no tiene fecha de vencimiento. Si toda la información que lo identifica o que puede identificarlo se elimina de la información sobre su salud, la información restante dejará de estar sujeta a esta autorización y podrá usarse o entregarse con otros fines.

Ninguna publicación ni presentación pública sobre la investigación descrita anteriormente revelarán su identidad sin que se haya obtenido otra autorización de parte suya.

## ¿Quién puede responder mis preguntas sobre esta investigación?

El investigador, Bijan Najafi, y/o la persona que él designe en su lugar intentarán responder todas sus preguntas. Si en algún momento tiene preguntas, quejas o preocupaciones, o si necesita comunicar una lesión relacionada con la investigación, puede hablar con un integrante del personal del estudio: Ivan Marin al número 713-798-7538 durante el día y fuera del horario de atención

Esta investigación está supervisada por un Comité de Revisión Institucional ("IRB"). El IRB es un grupo de personas que realizan revisiones de los estudios de investigación de manera independiente. Puede hablar con estas personas llamando al número (800) 562-4789 o a través del correo electrónico help@wirb.com si:

- Tiene preguntas, preocupaciones o quejas que no responde el equipo de la investigación.
- No recibe respuestas del equipo de la investigación.
- No puede localizar al equipo de la investigación.
- Quiere hablar con alguien más sobre la investigación.
- Tiene preguntas sobre sus derechos como sujeto de una investigación.

# ¿Qué sucede si sufro una lesión por participar en esta investigación?

Si sufre una lesión o se enferma por participar en esta investigación, llame de inmediato al médico del estudio, quien le brindará tratamiento médico de emergencia. Es posible que este tratamiento se le cobre a su seguro. El patrocinador pagará cualquier gasto que no cubra su póliza de seguro o el gobierno, siempre que la lesión no se haya debido a su afección o enfermedad subyacente y no la haya causado usted o algún otro tercero. Ni el patrocinador ni el médico del estudio disponen habitualmente de otro pago.

# ¿Pueden retirarme de esta investigación sin mi aprobación?

La persona a cargo de esta investigación puede retirarlo de la misma sin su aprobación. Los posibles motivos para el retiro incluyen lo siguiente:

- Es lo mejor para usted.
- Usted tiene un efecto secundario que requiere la interrupción de su participación en la investigación.
- Usted necesita un tratamiento que no se permite en esta investigación.
- El patrocinador cancela la investigación.
- Usted no puede cumplir con las citas programadas.

Le comunicaremos la información nueva que pueda afectar a su salud, a su bienestar o a su elección de seguir en esta investigación.

# ¿Qué sucede si acepto participar en esta investigación, pero cambio de opinión más adelante?

Si decide retirarse de esta investigación, comuníquese con el equipo de la investigación para que el investigador pueda hacer lo siguiente:

- Retirarlo del estudio.
- Comunicarle su retiro del estudio al médico que lo trata.
- Comunicar el motivo por el que usted decide no participar en el estudio de investigación.

Si decide retirarse de la investigación antes de tiempo, esta decisión puede implicar riesgos. Estos pueden incluir: Describir las consecuencias adversas.

#### ¿Se me pagará por participar en esta investigación?

Por la participación en esta investigación, se le puede pagar un total máximo de \$1,275. La compensación se distribuirá de la siguiente manera:

- Se le pagarán \$75 por cada visita que complete. Hay un total de 17 visitas.
- Se le entregará una tarjeta de débito llamada "ClinCard" el primer día de visita que tenga. Cada vez que complete una visita, el coordinador cargará \$75 a la tarjeta. Tenga en cuenta que para que la cantidad se cargue a la tarjeta pueden pasar hasta 72 horas. El coordinador de la investigación le dará algunas instrucciones e información útil sobre la tarjeta. Se le pedirá su número de seguro social para que el equipo de la investigación emita los pagos.
- El estudio de investigación también cubrirá sus gastos de estacionamiento o traslados para ir a las visitas de la investigación.

#### **DERECHOS DE LOS SUJETOS:**

Su firma en este formulario de consentimiento significa que ha recibido la información sobre este estudio y que acepta participar como voluntario en este estudio de investigación.

Recibirá una copia de este formulario firmado para que la guarde. Al firmar este formulario, usted no renuncia a ninguno de sus derechos. Incluso después de haber firmado este formulario, usted puede cambiar de opinión en cualquier momento. Comuníquese con el personal del estudio si decide dejar de participar en este estudio.

Si elige no participar en la investigación o si decide dejar de hacerlo más adelante, sus beneficios y servicios seguirán siendo los mismos que antes de que se analizara este estudio con usted. No perderá estos beneficios, servicios o derechos.

La firma de este formulario de consentimiento indica que usted lo ha leído (o que se lo han leído), que ha recibido respuestas satisfactorias a sus preguntas y que acepta voluntariamente participar en este estudio de investigación. Recibirá una copia de este formulario de consentimiento firmado.

Su firma documenta su permiso para que usted o la persona que se nombra a continuación participe en esta investigación.

| Firma del sujeto adulto capaz de dar el c | Fecha |
|----------------------------------------------------|-------------------|
| Nombre del sujeto (en letra de in | Fecha |
| (no se requiere si el sujeto dio personalmente su | a consentimiento) |
| Firma de la persona que obtiene el con | Fecha |
| Testigo (si corresponde) | Fecha |
| Traductor (si corresponde) | Fecha |
| , , | |
| BAYLOR COLLEGE OF MEDICINE & AFFILIATED HOSPITALS | |



BAYLOR COLLEGE OF MEDICINE & AFFILIATED HOSPITALS FOR HUMAN SUBJECT RESEARCH APPROVED BY THE DESIGNATED IRB: Western Institutional Review Board

APPROVED FROM: 12/03/2019

TO: 12/29/2020